CLINICAL TRIAL: NCT03029039
Title: Platelet-associated Inflammation in Severe Sepsis
Acronym: PlatISSep
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: 1608110; ID-RCB (Other: 2016-A01461-50)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Severe Sepsis
Keywords: Platelet; severe sepsis; inflammation; S. aureus; biomarkers
MeSH Terms: conditions — Sepsis; Inflammation; Staphylococcal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with severe sepsis: Blood samples will be collected at inclusion.
  Interventions: Other: Blood samples
- patients with inflammatory syndrome without sepsis: Blood samples will be collected at inclusion.
  Interventions: Other: Blood samples
- blood donor voluntary: Blood samples will be collected.
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples will be collected at inclusion.

SUMMARY:
Sepsis represents a serious public health issue characterized by a complex inflammatory response. In addition to their hemostatic role, platelets display inflammatory functions by secreting a variety of immunomodulatory factors and interacting with circulating immune cells. The investigators postulate that, in severe sepsis, platelets become activated and release amounts of different soluble inflammatory molecules that contribute to sepsis-associated inflammation. First, the investigators propose to assess whether severe sepsis impairs the ability of platelets to release soluble CD40L (sCD40L), an powerful platelet-derived immunomodulatory molecule, in ICU patients with S. aureus documented infection, ICU patients with documented infection involving other bacterial species, compared to ICU patients with inflammation of noninfectious origin and healthy blood donors. Then, the investigators wish to assess whether the bacterial species affects the release of platelet sCD40L and by an extensive screening of platelet soluble factors, the investigators propose to set up profiles of inflammatory molecules associated with the type of infection. Finally, the investigators will analyze platelets' activation state and their association with circulating immune, according to the type of infection. Therefore, this project is expected to assess to which extent the platelet inflammatory function is super-activated in severe sepsis and to identify new platelet-related biomarkers of sepsis.

ELIGIBILITY:
Inclusion criteria

Common inclusion criteria for ICU patients : Signed informed consent, Patient affiliated or entitled to a social security, aged over 18 years,

* Criteria for blood donor voluntary : to weigh more than 50 kg
* Criteria for severe sepsis group : Sepsis with failure of at least one organ, severe sepsis for less than 72 hours, sepsis with bacteria S. aureus, S. pneumoniae or E. coli.
* Criteria for uninfectious inflammatory syndrome group : patients operate since less than 24 hours of hip or knee surgery, Absence of systemic infection

Exclusion Criteria

* failure to participate at the study
* Patients with a aspirin treatment has continued throughout severe sepsis
* Patients with an appropriate antibiotic therapy for more than 72 hours
* Patients with a platelet transfusion in the week before inclusion or 72 hours after a surgical gesture or the occurrence of sepsis
* Patients with the platelet account is less than 30 000 per cubic millimeter the day of the sampling
* Patients with a severe sepsis who had a surgical gesture previous week the inclusion
* All clinical sequelae or biological at the selection
* pregnant woman
* Patients with a treatment by platelet aggregation has continued throughout severe sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with severe sepsis
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Comparison of proportion of CD40L between the 3 groups | 1 year
  Comparison of proportion of CD40L in Platelet-rich plasma (PRP) between the 3 groups by proteomics technique Luminex® stimulated by Thrombin Receptor Activator Peptide (TRAP)-6).

SECONDARY OUTCOMES:
Comparison of proportion of CD40L between patients with severe sepsis and blood donor voluntary | 1 year
  Comparison of proportion of CD40L in Platelet poor plasma (PPP) between patients with severe sepsis and blood donor voluntary by proteomics technique Luminex® stimulated by Thrombin Receptor Activator Peptide (TRAP)-6).
Comparison of proportion of CD40Lbetween patients with severe sepsis and patients with inflammatory syndrome without sepsis | 1 year
  Comparison of proportion of CD40L in Platelet-rich plasma (PRP) between patients with severe sepsis and patients with inflammatory syndrome without sepsis by proteomics technique Luminex® stimulated by Thrombin Receptor Activator Peptide (TRAP)-6).
Proportion of CD40L | 1 year
  Proportion of CD40L of patients with severe sepsis according to the different infection (S. aureus , S. pneumoniae, E. coli)

CONTACTS AND LOCATIONS:
Overall Officials: Phillipe BERTHELOT, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No